CLINICAL TRIAL: NCT05140538
Title: A New Domiciliary Oral Care Protocol for the Management of Dental Erosion in Rugby Players: A Randomized Clinical Trial
Brief Title: A New Protocol for the Management of Dental Erosion in Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-RUGBY
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Dental Erosion
Keywords: enamel remineralization
MeSH Terms: conditions — Tooth Erosion | interventions — Toothpastes; Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): SRP + Biorepair Total Protective Repair toothpaste for home oral hygiene twice a day
  Interventions: Other: SRP + toothpaste
- Group 2 (Experimental): SRP + Biorepair Total Protective Repair toothpaste + Biorepair mouthwash (3 in 1) for home oral hygiene twice a day
  Interventions: Other: SRP + toothpaste + mouthwash

INTERVENTIONS:
Other: SRP + toothpaste + mouthwash — Use of domiciliary products twice a day
  Arms: Group 2
Other: SRP + toothpaste — Use of domiciliary products twice a day
  Arms: Group 1

SUMMARY:
The aim of the present study is to provide a new domiciliary oral care treatment for enamel remineralization in rugby players patients using mouthguards. Patients selected for the study will be randomly divided and allocated in two groups according to the treatment:

* Group 1: scaling and root planing (SRP) + Biorepair Total Protective Repair toothpaste for home oral hygiene twice a day
* Group 2: scaling and root planing (SRP) + Biorepair Total Protective Repair toothpaste + Biorepair mouthwash (3 in 1) for home oral hygiene twice a day

Patients will be given instructions for the cleaning of their mouthguards. The periodontal evaluation will be conducted before SRP, after 15, 30 and 90 days. The periodontal indices collected will be: PI, BoP, Schiff Air Index, BEWE index and dental sensitivity (VAS scale).

DETAILED DESCRIPTION:
The aim of the present study is to provide a new domiciliary oral care treatment for enamel remineralization in rugby players patients using mouthguards and to prevent further worsening of dental erosion. Patients selected for the study will sign the informed consent and will be randomly divided and allocated into two groups:

* Group 1: SRP + Biorepair Total Protective Repair toothpaste for home oral hygiene twice a day
* Group 2: SRP + Biorepair Total Protective Repair toothpaste + Biorepair mouthwash (3 in 1) for home oral hygiene twice a day

Patients will be given instructions for the cleaning of their mouthguards. The periodontal evaluation will be conducted before SRP, after 15, 30 and 90 days. The periodontal indices collected will be: PI, BoP, Schiff Air Index, BEWE index and dental sensitivity (VAS scale).

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate to the study
* Rugby players

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients suffering from neurological disorders
* Patients suffering from psychological disorders
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in BOP - Bleeding on Probing (percentage) | Study begin, 1 and 3 months
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 4 sites (mesial, distal, vestibular, palatal/lingual).
Change in Schiff Air Index - Dental sensitivity test | Study begin and after 15, 30 and 90 days.
  Scoring criteria:
  0: the subject did not respond to air blasting;
  1. the subject responded to air blasting;
  2. the subject responded to air blasting and requested discontinuation;
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change of the BEWE Index - Basic Erosive Wear Examination (Barlet et al., 2008) | Study begin and after 15, 30 and 90 days.
  Scoring criteria:
  0: no erosive tooth wear;
  1. initial loss of surface texture;
  2. distinct defect, hard tissue loss < 50% of the surface area;
  3. hard tissue loss ≥ 50% of the surface area.
Change in PI - Plaque Index (percentage) | Study begin and after 15, 30 and 90 days.
  Evaluation of the presence of plaque with a disclosing agent on the 4 surfaces of teeth on the total amount of dental surfaces multiplied per 100.
Dental sensitivity | Study begin and after 15, 30 and 90 days.
  Assessment of dental sensitivity with a VAS scale (score: from 1 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.